CLINICAL TRIAL: NCT00320749
Title: A Dose Escalating (Phase I) Study Looking at the Biomodulation of Capecitabine by Docetaxel and Gemcitabine in Patients With Advanced Pancreas Cancer
Brief Title: Capecitabine, Docetaxel and Gemcitabine in Patients With Advanced Pancreas Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tony Bekaii-Saab (Other)
Collaborators: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor-Investigator, Tony Bekaii-Saab, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-05058
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Results first posted 2015-10-19 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-05

CONDITIONS: Pancreatic Cancer
Keywords: Advanced Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine; Docetaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- capecitabine, docetaxel, gemcitabine (Experimental): Dose escalation study of mGTX using three dose levels (DL1-3). Patients received docetaxel on days 1 and 8, gemcitabine on days 8 and 15, and capcitabine on days 8 through 21. Gemcitabine fixed dose at 750 mg/m2 over 75 min, capecitabine twice daily and escalated from 500 to 650 mg/m2 at DL2 and docetaxel increased from 30 to 36 mg/m2 at DL3.
  Interventions: Drug: Capecitabine; Drug: Docetaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Capecitabine — Will be give on days 8-21
  Other Names: Xeloda
Drug: Docetaxel — Will be given on days 1 and 8,
  Other Names: Taxotere
Drug: Gemcitabine — A fixed dose rate will be give on days 8 and 15.
  Other Names: Gemzar

SUMMARY:
The primary purpose of this study is to define the maximum tolerated dose of combination docetaxel, gemcitabine, and capecitabine in patients with pancreatic cancer. Adverse effects will be measured in study participants. In addition, researchers will assess data about preliminary efficacy in patients with this treatment approach.

DETAILED DESCRIPTION:
Rationale: Single agent gemcitabine is considered standard care for patients with advanced pancreatic cancer. However, better treatments offering improved outcomes are needed for people with this disease. The combination of docetaxel and capecitabine has shown significant and broad clinical activity in a variety of tumors. Laboratory research on the combination of capecitabine, docetaxel, and gemcitabine indicates synergistic action against tumor cells. The current study will test this combination in patients. The drug administration schedule in this study is aimed at maximizing the potential of activation of capecitabine by both docetaxel and gemcitabine.

Treatment: Study participants will be given docetaxel, gemcitabine, and capecitabine. All study drugs will be administered through intravenous infusions in three week cycles. Docetaxel will be given on days 1 and 8, gemcitabine on days 8 and 15, and capecitabine on days 8 through 21. This schedule will be followed by 1 week of rest without administration of study drugs. Since the primary goal of this study is to identify the maximum tolerated dose of the study drugs in combination, patients who enroll in the beginning of the study will receive lower amounts of the study drugs compared to patients who enroll later in the study. Several tests and exams will be given throughout the study to closely monitor patients.

ELIGIBILITY:
Inclusion Criteria:

* adenocarcinoma of the pancreas
* no prior chemo except adjuvant
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* peripheral neuropathy </= Gr. 1

Exclusion Criteria:

* Pregnant/lactating females
* Uncontrolled heart disease, diabetes, psychiatric disorder
* Therapeutic doses of Warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2005-12; Primary Completion 2008-10 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanios Saab, Principal Investigator — Ohio State University; Tanios Saab, M.D., Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - The University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Ohio State University, Columbus, Ohio

REFERENCES:
- [Result] Hill ME, Li X, Kim S, Campbell A, Culler K, Bloomston M, Zalupski M, Hejna G, Bekaii-Saab T. A phase I study of the biomodulation of capecitabine by docetaxel and gemcitabine (mGTX) in previously untreated patients with metastatic adenocarcinoma of the pancreas. Cancer Chemother Pharmacol. 2011 Mar;67(3):511-7. doi: 10.1007/s00280-010-1348-3. Epub 2010 May 12. PMID 20461379
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled into the study between December 2005 and February 2008.
Pre-assignment Details: Patients had histologically or cytologically confirmed metastatic pancreatic adenocarcinoma and measurable disease per RECIST criteria.
Groups:
- Dose Level 1: Docetaxel at 30 mg/m2 on days 1 and 8, Gemcitabine at 750 mg/m2 (over 75 minutes) on days 8 and 15 and capecitabine at 500 mg/m2/12 hours on days 8-21
- Dose Level 2: Docetaxel at 30 mg/m2 on days 1 and 8, Gemcitabine at 750 mg/m2 (over 75 minutes) on days 8 and 15 and capecitabine at 625 mg/m2/12 hours on days 8-21
- Dose Level 3: Docetaxel at 36 mg/m2 on days 1 and 8, Gemcitabine at 750 mg/m2 (over 75 minutes) on days 8 and 15 and capecitabine at 625 mg/m2/12 hours on days 8-21
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Started | 3 | 8 | 10
Completed | 3 | 6 | 1
Not Completed | 0 | 2 | 9

BASELINE CHARACTERISTICS:
Groups:
- Capecitabine, Gemcitabine and Docetaxel: Docetaxel i.v. over 30 min on days 1 and 8; Capecitabine p.o. in split doses bid on days 8-21, Gemcitabine i.v. over 75 min on days 8 and 15.
Arm/Group | Capecitabine, Gemcitabine and Docetaxel
Number analyzed (Participants) | 21
Age, Continuous [Mean (Full Range); unit: years] | 59 [48 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 21
Eastern Cooperative Oncology Group (ECOG) [Number; unit: patients]
  ECOG 0 (Fully Active) | 4
  ECOG 1 (Restricted physical activity) | 17

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: MTD will be the dose at which 1 or fewer patients (≤ 1/6) experiences a DLT during the first or second cycle with the next higher dose having at least 2/3 or 2/6 patients experiencing Dose Limiting Toxicities (DLT).
Time Frame: Weekly up to 24 weeks
Measure: Number; unit: mg/m^2
Groups:
- Capecitabine, Docetaxel, Gemcitabine: Dose escalation study of mGTX using three dose levels (DL1-3). Patients received docetaxel on days 1 and 8, gemcitabine on days 8 and 15, and capecitabine on days 8 through 21. Gemcitabine fixed dose at 750 mg/m2 over 75 min, capecitabine twice daily and escalated from 500 to 650 mg/m2 at DL2 and docetaxel increased from 30 to 36 mg/m2 at DL3.
  Capecitabine: Will be give on days 8-21
  Docetaxel: Will be given on days 1 and 8,
  Gemcitabine: A fixed dose rate will be give on days 8 and 15.
Arm/Group | Capecitabine, Docetaxel, Gemcitabine
Number analyzed (Participants) | 21
mg/m^2
  docetaxel | 36
  gemcitabine | 750
  capecitabine | 625

2. Secondary Outcome: Common Toxicities
Description: The NCI Common Terminology Criteria for Adverse Events version 3.0 was used for adverse event reporting and toxicity grading.
Time Frame: Weekly up to 24 weeks
Population: grade 3 and grade 4 toxicities according to National Cancer Institute [NCI] Common Toxicity Criteria for Adverse Events [CTCAE], Version 3.0
Measure: Number; unit: percent of patients
Groups:
- Capecitabine, Docetaxel, Gemcitabine: Dose escalation study of mGTX using three dose levels (DL1-3). Patients received docetaxel on days 1 and 8, gemcitabine on days 8 and 15, and capecitabine on days 8 through 21. Gemcitabine fixed dose at 750 mg/m2 over 75 min, capecitabine twice daily and escalated from 500 to 650 mg/m2 at DL2 and docetaxel increased from 30 to 36 mg/m2 at DL3.
Arm/Group | Capecitabine, Docetaxel, Gemcitabine
Number analyzed (Participants) | 21
percent of patients
  leukopenia | 29
  neutropenia | 29
  fatigue | 25

3. Secondary Outcome: Therapeutic Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: every 8 weeks, up to 24 weeks
Population: 3 patients were non-evaluable for response or progression free survival as they withdrew consent after cycle 1 of therapy.
Measure: Number; unit: percent of patients
Arm/Group | Capecitabine, Docetaxel, Gemcitabine
Number analyzed (Participants) | 18
percent of patients
  Partial Response | 11
  Complete Response | 0
  Stable Disease | 72

ADVERSE EVENTS:
Arm/Group | Capecitabine, Docetaxel, Gemcitabine
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 21/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capecitabine, Docetaxel, Gemcitabine (N=21)
Leukopenia (Blood and lymphatic system disorders) | 14 (14)
Neutropenia (Blood and lymphatic system disorders) | 11 (11)
Anemia (Blood and lymphatic system disorders) | 10 (10)
Thrombocytopenia (Injury, poisoning and procedural complications) | 10 (10)
Fatigue (General disorders) | 18 (18)
Nausea (Gastrointestinal disorders) | 16 (16)
Diarrhea (Gastrointestinal disorders) | 16 (16)
Alopecia (Skin and subcutaneous tissue disorders) | 13 (13)
Neuropathy (Nervous system disorders) | 11 (11)
Vomiting (Gastrointestinal disorders) | 8 (8)
Mucositis (Gastrointestinal disorders) | 7 (7)
Transaminitis (Infections and infestations) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes